CLINICAL TRIAL: NCT05060861
Title: Safety, Efficacy and Immunogenicity of Chadox1 Ncov-19 Vaccine: Rapid Systematic Review and Meta Analysis
Brief Title: Safety, Efficacy of Chadox1 Ncov-19 Vaccine: Rapid Systematic Review and Meta Analysis
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Aliae AR Mohamed Hussein, Professor of Pulmonology, Assiut University
Other Study IDs: Assiut19
Record Dates: First submitted 2021-09-18; First posted 2021-09-29 (Actual); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: ChAdOx1 nCoV-19 Vaccine
Keywords: safety; efficacy; immunogenicity; COVID-19 vaccine
MeSH Terms: interventions — ChAdOx1 nCoV-19

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: ChAdOx1 nCoV-19 vaccine — covid-19 vaccine

SUMMARY:
Since the beginning of COVID-19 pandemic, a safe and effective vaccine against infection and development of acute respiratory syndrome coronavirus 2 (SARS-CoV-2) is needed control of the wide spread of COVID-19 and reduce death rates throughout the world. Many clinical trials investigated the immunogenicity of different proposed vaccine including the first distributed vaccine; the ChAdOx1 nCoV-19 vaccine and there is a need to analyze the results of published clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* Participant who received 2 doses of ChAdOx1 nCoV-19 vaccine

Exclusion Criteria:

* non vaccinated person

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Participants aged 18 years and older vaccinated by 2 doses of ChAdOx1 nCoV-19 vaccine
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2021-08-30 (Actual); Study Completion 2021-10-30 (Estimated)

PRIMARY OUTCOMES:
To evaluate the safety and efficacy of the ChAdOx1 nCoV-19 vaccine in a pooled interim analysis | up to one year
  the frequency of breakthrough COVID-19 infection

CONTACTS AND LOCATIONS:
Locations (1):
- Aliae AR Mohamed-Hussein, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
upon reasonable request